CLINICAL TRIAL: NCT03464773
Title: Optimizing the Management of Pain and Irritability of Unknown Origin (PIUO) in Children With Severe Neurological Impairment
Brief Title: Pain and Irritability in Non-Verbal Children
Acronym: PIUO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Calgary (Other); University of Ottawa (Other); Provincial Health Services Authority British Columbia (Other); Alberta Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Harold Siden, Dr., University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H16-03288
Record Dates: First submitted 2018-01-25; First posted 2018-03-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pain; Neuropathic Pain; Irritability
MeSH Terms: conditions — Pain; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathway (Other): The PIUO Pathway is implemented by clinicians (MD and RN) with expertise in treating pain in children. Each participant proceeds through the PIUO Pathway as long as their pain persists, but will exit the PIUO Pathway at any stage in case their pain is resolved. The Pathway has two steps: Step 1 is a thorough history and patient evaluation, including directed testing. Step 2 is a series of screening tests to further explore any potential underlying disease or injury not apparent based on history and physical examination.
  Interventions: Other: PIUO Pathway
- Waitlist (No Intervention): Participants randomized to the Waitlist will cross over to the Pathway after 8 weeks.

INTERVENTIONS:
Other: PIUO Pathway — See arm descriptions
  Arms: Pathway

SUMMARY:
Children born with severe brain-based developmental disabilities frequently experience persistent unexplained periods of pain and irritability, often compounded by a limited capacity to communicate their distress. The investigators call this entity Pain and Irritability of Unknown Origin (PIUO). The investigators have designed a systematic approach, called the PIUO Pathway, to address the management of these children's pain and irritability with the goals of reducing pain symptoms, improving the day-to-day lives of the child and family, and simplifying treatment options for clinicians.

DETAILED DESCRIPTION:
The purpose of this project is to develop, test, and disseminate an approach to reducing and resolving pain in children with developmental brain disorders, specifically those with severe neurological impairments (SNI). It focuses on the problem of ongoing, unexplained, and difficult-to-treat pain and irritability that many children with SNI, and their families, experience over time. The goal is to improve the assessment and treatment of pain and irritability in children diagnosed with complex health conditions and multiple disabilities, who have limited communication and cognition.

The plan is to evaluate the effectiveness of an integrated clinical pathway (i.e. a sequential order of standardized evaluation steps) for managing unexplained pain and irritability in these vulnerable children.

BACKGROUND Pain is the most common symptom reported by the parents and caregivers of children with SNI, however, pain is notoriously difficult to identify, and therefore treat, in non-verbal children because their signals of distress are ambiguous and hard to decode. Typical distress behaviours include crying, tears, facial grimace, limb withdrawal, arching, hypertonicity, and decreased sleep. More mobile children may curl up into a ball, fling their arms or legs, or engage in self-injurious behaviour; conversely they may display decreased activity.

Children with SNI may experience nociceptive-inflammatory pain as a result of their specific medical condition (e.g. joint contractures) or from many procedures that they experience (e.g. injections). Often, however, it is not clear what underlies the pain behavior. Parents are experts in identifying pain behaviours in their own child, but consider their interpretation to be a complex and uncertain process. As well, while pain behaviours can be described by clinicians and parents, the behaviours themselves are subjective, ambiguous, and can reflect a variety of problems in addition to pain. Unless an obvious nociceptive-inflammatory trigger such as an injury is witnessed, parents and clinicians find it very difficult to ascribe all of the pain-like behaviours observed in children with SNI to pain as defined by the International Association for the Study of Pain (IASP). In this context, the term "pain" does not serve as a descriptive label. Therefore, the investigators describe pain behaviour episodes using a less deterministic term, "pain and irritability," acknowledging that the behaviour is certainly negative in the eyes of the witnessing caregiver. The team has defined this entity as Pain and Irritability of Unknown Origin (PIUO).

HYPOTHESIS The overall hypothesis is that children participating in the PIUO Pathway will experience improvement or resolution of PIUO from baseline to post-study, compared to children receiving treatment as usual while on the waitlist.

The goal is to improve PIUO beyond what has been undertaken by the child's usual clinical teams. The primary outcome is improved pain control for non-verbal children with SNI as shown in a reduction of pain and irritability episodes and their severity. Secondary outcomes include decreased pain severity; improved family quality of life and ease of implementation of the PIUO Pathway for clinicians.

STUDY DESIGN Interventions for resolving PIUO are time- and resource-intensive. They require a focused approach to assessing all the underlying possibilities for the PIUO and addressing each potential source of pain one at a time. Tackling PIUO requires systematic, comprehensive, process-oriented thinking applied by an interdisciplinary team with flexibility in terms of approach and time. There have been recommendations in the literature about how to approach the problem of PIUO in children with SNI, but these recommendations have never been subjected to systemic evaluation as complex interventions, for example by following an integrated clinical pathway.

Integrated clinical pathways (also called "care pathways" or "critical pathways") are structured, sequenced approaches guiding the delivery of healthcare, often with a multidisciplinary perspective. They provide algorithms to be followed in the assessment and treatment of conditions, but are not intended to be rigidly followed; instead, integrated clinical pathways delineate a foundation for a clinician's approach to a complex problem, thereby avoiding inefficiencies in evaluation or resource use. Integrated clinical pathways are a form of Complex Interventions and have been developed for sickle cell pain, childhood asthma, appendicitis, autoimmune conditions, in-born errors of metabolism, and cerebrospinal fluid shunt management. Despite their complexity, integrated clinical pathways are appropriate interventions for evaluation by Randomized Controlled Trial (RCT). RCTs of integrated clinical pathways have been proposed and/or completed for complex, multi-factorial patient problems including lung disease, heart failure, gastrointestinal surgery, stroke, and hip fractures.

In this study, the investigators will use a waitlist-controlled RCT design, with 120 children randomized to PIUO Pathway or waitlist (standard care) treatment arms. This design was chosen strategically, with consideration of both the special pediatric population being studied and the ethical inappropriateness of randomly assigning children to a placebo group when pain is the target condition.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 18 years with SNI (from any cause) with unexplained pain and irritability and whose cognitive or communication impairments prevent determination of pain location, cause, and type will be eligible to participate.
* Eligible children will have cognitive impairment or be non-verbal and have severe levels of disability equivalent to Gross Motor Functional Classification System (GMFCS) scores of 3, 4 or 5.
* Eligible children will score >3 on two scales administered via an Eligibility Screening that measures persistence and distress level the child is experiencing as well as identifies the type of pain and irritability as PIUO - with no obvious cause or explanation. The score of >3 on the scale measuring pain persistence and distress level confirms that the child is experiencing pain and irritability more than "a little" on "some days".
* Parents should have sufficient English/French language skill, or have access to assistance, to participate in the clinic visits and complete survey tools.

Exclusion Criteria:

* Children not within the specified age range
* Children with communication capabilities and cognitive development to localize their pain
* Children that have an explained and treatable cause of pain and irritability.
* Parents who do not speak one of Canada's two official languages (English or French)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Reduction of pain severity of children on the pathway | Week 10
  Number of participants whose pain scores rank in the lower pain categories (category A or B) as compared to the proportion of those on the waitlist group, measured by the parent-reported Pain Survey.

SECONDARY OUTCOMES:
Identification of causes of pain and irritability of unknown origin in non-verbal children | End of Pathway (up to 8 months post-baseline)
  Number of children with known causes of pain and irritability at end of pathway
Decreased pain & irritability scores for children over time | Baseline and End of Pathway (up to 8 months post-baseline)
  Pain Survey (baseline score compared to End of Pathway score)
Improvement in parent fatigue levels | Baseline and End of Pathway (up to 8 months post-baseline)
  Parent-reported reduction in fatigue levels on the Patient-Reported Outcomes Measurement Information System (PROMIS-57: Fatigue 8a subscale Max. 40 to Min. 8- higher values worse) from baseline fatigue score compared to End of Pathway score
Recorded time commitment for clinical team to implement PIUO Pathway | Baseline and End of Pathway (up to 8 months post-baseline)
  Average hours of clinical time for MD + RD involved to complete the study per patient
Benefit ranking of ongoing communication with study research nurse | End of Pathway (up to 8 months post-baseline)
  Number of parents rating the communication with the nurse as "valuable" as per the Family feedback form.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Siden, MD, Principal Investigator — BC Children's Hospital Research Institute
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siden HB, Carleton BC, Oberlander TF. Physician variability in treating pain and irritability of unknown origin in children with severe neurological impairment. Pain Res Manag. 2013 Sep-Oct;18(5):243-8. doi: 10.1155/2013/193937. Epub 2013 Jul 24. PMID 23885348
- See also: Study website — http://www.paindetectives.org

DOCUMENTS (1):
  • Study Protocol (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03464773/Prot_002.pdf